CLINICAL TRIAL: NCT00670007
Title: An Open-label, Non-controlled, Multicenter, Multinational Study to Evaluate the Efficacy and Safety of Zemaira® Administration in Chronic Augmentation and Maintenance Therapy in Subjects With Emphysema Due to alpha1-proteinase Inhibitor Deficiency Who Completed Clinical Study CE1226_4001
Brief Title: Extension Study of Zemaira® i.v. Administration in Subjects With Emphysema Due to alpha1-proteinase Inhibitor Deficiency.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE1226_3001; 1466 (Other: CSL Behring); 2007-007129-38 (EudraCT Number)
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Results first posted 2016-07-12 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-07

CONDITIONS: Emphysema; Alpha 1-proteinase Inhibitor Deficiency
Keywords: Alpha1-proteinase inhibitor deficiency; Chronic augmentation and maintenance therapy; Emphysema; Emphysema due to Alpha 1-proteinase inhibitor deficiency
MeSH Terms: conditions — Emphysema; alpha 1-Antitrypsin Deficiency | interventions — alpha 1-Antitrypsin; Respreeza

ARMS (1):
- Zemaira® (Experimental)
  Interventions: Biological: Alpha1- proteinase inhibitor [human]

INTERVENTIONS:
Biological: Alpha1- proteinase inhibitor [human] — Lyophilized preparation of 60 mg/kg body weight intravenously once per week
  Other Names: Zemaira®; Respreeza®

SUMMARY:
This study is a continuation of the placebo-controlled study CE1226_4001 (NCT00261833) to evaluate the efficacy and safety of Zemaira® intravenous (i.v). administration in subjects with emphysema due to alpha1-proteinase inhibitor deficiency. The long-term verification of a disease-modifying benefit of Zemaira® on the progression of emphysema will be assessed by volume-adjusted lung density, measured yearly by computed tomography (CT).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed the 2-year treatment and observation period in the Phase 3/4 Zemaira® CE1226_4001 study (NCT00261833) and are willing to sign informed consent
* Males, and non-pregnant, non-lactating females, whose screening pregnancy test is negative and who are using contraceptive methods deemed reliable by the investigator

Exclusion Criteria:

* Individuals residing in the US
* Current evidence of alcohol abuse or abuse of drugs such as barbiturates, benzodiazepines, amphetamines, cocaine, opioids, and cannabinoids
* History of allergy, anaphylactic reaction, or severe systemic response to human plasma derived products, or known mannitol hypersensitivity, or history of prior adverse reaction to mannitol
* Current tobacco smoker (smoking must be discontinued for at least 6 months prior to study participation)
* Conditions or behaviors that interfere with attending scheduled study visits in the opinion of the investigator
* History of non-compliance
* Administration of any other experimental new drug or participation in an investigation of a marketed product
* Inability to perform necessary study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2008-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Clinical R&D, Study Director — CSL Behring
Locations (21):
- Australia (5):
  - Study Site, Adelaide, South Australia
  - Study Site, Fitzroy, Victoria
  - Study Site, Darlinghurst
  - Study Site, Nedlands
  - Study Site, New Lambton
- Canada (3):
  - Study Site, Vancouver, British Columbia
  - Study Site, Halifax, Nova Scotia
  - Study Site, Toronto, Ontario
- Study Site, Praha 4 - Krc, Czechia
- Denmark (2):
  - Study Site, Arhus C
  - Study Site, Hellerup
- Study Site, Tartu, Estonia
- Study Site, Oulu, Finland
- Germany (3):
  - Study Site, Essen
  - Study Site, Heidelberg
  - Study Site, Nuremberg
- Study Site, Dublin, Ireland
- Poland (2):
  - Study Site, Krakow
  - Study Site, Warsaw
- Study Site, Bucharest, Romania
- Study Site, Malmo, Sweden

REFERENCES:
- [Derived] Greulich T, Chlumsky J, Wencker M, Vit O, Fries M, Chung T, Shebl A, Vogelmeier C, Chapman KR, McElvaney NG; RAPID Trial Group. Safety of biweekly alpha1-antitrypsin treatment in the RAPID programme. Eur Respir J. 2018 Nov 29;52(5):1800897. doi: 10.1183/13993003.00897-2018. Print 2018 Nov. PMID 30237305
- [Derived] McElvaney NG, Burdon J, Holmes M, Glanville A, Wark PA, Thompson PJ, Hernandez P, Chlumsky J, Teschler H, Ficker JH, Seersholm N, Altraja A, Makitaro R, Chorostowska-Wynimko J, Sanak M, Stoicescu PI, Piitulainen E, Vit O, Wencker M, Tortorici MA, Fries M, Edelman JM, Chapman KR; RAPID Extension Trial Group. Long-term efficacy and safety of alpha1 proteinase inhibitor treatment for emphysema caused by severe alpha1 antitrypsin deficiency: an open-label extension trial (RAPID-OLE). Lancet Respir Med. 2017 Jan;5(1):51-60. doi: 10.1016/S2213-2600(16)30430-1. Epub 2016 Dec 2. PMID 27916480
- [Derived] Chapman KR, Burdon JG, Piitulainen E, Sandhaus RA, Seersholm N, Stocks JM, Stoel BC, Huang L, Yao Z, Edelman JM, McElvaney NG; RAPID Trial Study Group. Intravenous augmentation treatment and lung density in severe alpha1 antitrypsin deficiency (RAPID): a randomised, double-blind, placebo-controlled trial. Lancet. 2015 Jul 25;386(9991):360-8. doi: 10.1016/S0140-6736(15)60860-1. Epub 2015 May 27. PMID 26026936

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted at 22 centers in Europe, Canada, and Australia.
  Alpha1-proteinase inhibitor (A1-PI) deficient individuals with emphysema, who had completed the 2-year treatment and observation periods in study CE1226_4001, except those participating in the USA, were invited to participate in study CE1226_3001.
Pre-assignment Details: Subjects who had participated in the CE1226_4001 study, met the inclusion and exclusion criteria, and signed the informed consent were included in study CE1226_3001.
Groups:
- Zemaira®: Alpha1- proteinase inhibitor [human]: Lyophilized preparation of 60 mg/kg body weight administered intravenously once per week
Period: Overall Study
Arm/Group | Zemaira®
Started | 140
Completed | 131
Not Completed | 9
Not completed — Drug abuse | 1
Not completed — Lung transplant | 1
Not completed — Travel/Vacation | 1
Not completed — Adverse event, serious fatal | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Zemaira®
Number analyzed (Participants) | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 130
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 79
Region of Enrollment [Number; unit: participants]
  Canada | 25
  Sweden | 17
  Czech Republic | 2
  Romania | 1
  Ireland | 19
  Finland | 3
  Poland | 4
  Denmark | 35
  Australia | 17
  Germany | 15
  Estonia | 2

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change of Adjusted Lung Density
Description: As measured by centralized, standardized computer tomographic (CT) lung densitometry. CT scans were acquired at 2 inspiration states: TLC (Total Lung Capacity; ie, full inspiration) and FRC (Functional Residual Capacity; ie, full expiration). Results were adjusted for total lung volume and are presented as point estimates for the average rate of decline in the early start and delayed start subgroups from a linear random regression model with country, inspiration state (only for 'TLC and FRC state'), time (time elapsed since Day 1 [CE1226_4001]), treatment and treatment by time interaction as fixed effects and subject and subject by time interaction as random coefficients.
Time Frame: Up to 2 years
Population: Intention-to-treat (ITT) population. Subjects may not have been included in all efficacy analyses because of missing efficacy assessments.
Measure: Least Squares Mean (Standard Error); unit: g/L per year
Groups:
- Zemaira® (Early Start): Those subjects who had already been allocated to receive Zemaira® treatment during study CE1226_4001 represent the Early Start group. This group had received up to 4 years of continuous therapy at the end of study CE1226_3001.
- Zemaira® (Delayed Start): Subjects who received placebo in study CE1226_4001 and only began to receive Zemaira® treatment upon entry into study CE1226_3001 represent the Delayed Start group. This group had a maximal exposure of 2 years at the end of study CE1226_3001.
Arm/Group | Zemaira® (Early Start) | Zemaira® (Delayed Start)
Number analyzed (Participants) | 75 | 64
g/L per year
  TLC + FRC combined | -1.632 (0.2824) | -1.352 (0.2961)
  TLC | -1.627 (0.2743) | -1.256 (0.2891)
  FRC | -1.658 (0.3186) | -1.482 (0.3346)
Statistical Analysis 1: Comparison: Zemaira® (Early Start) vs Zemaira® (Delayed Start); Analysis of the annual rate of change in lung density (for TLC + FRC combined) was a linear random regression model with country, inspiration state, time since Day 1 [CE1226_4001], and treatment-by time interaction as fixed effects and subject and subject-by-time interaction as random coefficients at a 1-sided significance level of 0.025; Test type: Superiority or Other; p = 0.752, Regression, Linear — A 1-sided P-value < 0.025 and a positive estimate of the treatment difference Early Start minus Delayed Start (ie, the lower bound of the 95% confidence interval [CI] being > zero) will indicate superiority of Early Start compared with Delayed Start; Difference in lung density(adjusted P15) = -0.279, 95% CI 2-sided [-1.089 to 0.530]
Statistical Analysis 2: Comparison: Zemaira® (Early Start) vs Zemaira® (Delayed Start); Analysis of the annual rate of change in lung density (for TLC) was a linear random regression model with country, time since Day 1 [CE1226_4001], and treatment-by-time interaction as fixed effects and subject and subject-by-time interaction as random coefficients at a 1-sided significance level of 0.025; Test type: Superiority or Other; p = 0.823, Regression, Linear — A 1-sided P-value < 0.025 and a positive estimate of the treatment difference Early Start minus Delayed Start (ie, the lower bound of the 95% CI being > zero) will indicate superiority of Early Start compared with Delayed Start; Difference in lung density(adjusted P15) = -0.371, 95% CI 2-sided [-1.159 to 0.417]
Statistical Analysis 3: Comparison: Zemaira® (Early Start) vs Zemaira® (Delayed Start); Analysis of the annual rate of change in lung density (for FRC) was a linear random regression model with country, time since Day 1 [CE1226_4001], and treatment-by-time interaction as fixed effects and subject and subject-by-time interaction as random coefficients at a 1-sided significance level of 0.025; Test type: Superiority or Other; p = 0.648, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Difference in lung density(adjusted P15) = -0.176, 95% CI 2-sided [-1.09 to 0.738]

2. Secondary Outcome: Absolute Change in Adjusted Lung Density
Description: Absolute change from baseline to 2 years as measured by centralized, standardized CT lung densitometry. CT scans were acquired at 2 inspiration states: TLC (ie, full inspiration) and FRC (ie, full expiration). Results were adjusted for total lung volume and are presented as point estimates for the average absolute change in the early start and delayed start subgroups from an analysis of covariance (ANCOVA) model with country, treatment, and baseline lung density as fixed effects and inspiration state as a repeated random effect. The baseline is the last assessment from the preceding study CE1226_4001.
Time Frame: From baseline to 2 years
Population: ITT population. Subjects may not have been included in all efficacy analyses because of missing efficacy assessments.
Measure: Least Squares Mean (Standard Error); unit: g/L
Arm/Group | Zemaira® (Early Start) | Zemaira® (Delayed Start)
Number analyzed (Participants) | 64 | 60
g/L
  TLC + FRC combined, n = 64, 60 | -3.031 (0.5888) | -2.502 (0.6142)
  TLC, n = 64, 59 | -2.971 (0.5826) | -2.485 (0.6142)
  FRC, n = 64, 60 | -2.934 (0.6671) | -2.953 (0.6993)
Statistical Analysis 1: Comparison: Zemaira® (Early Start) vs Zemaira® (Delayed Start); Analysis of the change in lung density (for TLC + FRC combined) from baseline to 2 years was analyzed using an ANCOVA model with country, treatment, and baseline lung density as fixed effects and inspiration state as a repeated random effect; Test type: Superiority or Other; p = 0.526, ANCOVA — Two-sided P-value; Difference in lung density(adjusted P15) = -0.530, 95% CI 2-sided [-2.179 to 1.120]
Statistical Analysis 2: Comparison: Zemaira® (Early Start) vs Zemaira® (Delayed Start); Analysis of the change in lung density (for TLC) from baseline to 2 years was analyzed using an ANCOVA model with country, treatment, and baseline lung density as fixed effects; Test type: Superiority or Other; p = 0.558, ANCOVA — Two-sided P-value; Difference in lung density(adjusted P15) = -0.486, 95% CI 2-sided [-2.126 to 1.154]
Statistical Analysis 3: Comparison: Zemaira® (Early Start) vs Zemaira® (Delayed Start); Analysis of the change in lung density (for FRC) from baseline to 2 years was analyzed using an ANCOVA model with country, treatment, and baseline lung density as fixed effects; Test type: Superiority or Other; p = 0.984, ANCOVA — Two-sided P-value; Difference in lung density(adjusted P15) = 0.019, 95% CI 2-sided [-1.858 to 1.895]

3. Secondary Outcome: Percent Change in Adjusted Lung Density
Description: Percent change from baseline to 2 years as measured by centralized, standardized CT lung densitometry. CT scans were acquired at 2 inspiration states: TLC (ie, full inspiration) and FRC (ie, full expiration). Results were adjusted for total lung volume and are presented as point estimates for the average percent change in the early start and delayed start subgroups from an analysis of covariance (ANCOVA) model with country, treatment, and baseline lung density as fixed effects and inspiration state as a repeated random effect. The baseline is the last assessment from the preceding study CE1226_4001.
Time Frame: From baseline to 2 years
Population: ITT population. Subjects may not have been included in all efficacy analyses because of missing efficacy assessments.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Zemaira® (Early Start) | Zemaira® (Delayed Start)
Number analyzed (Participants) | 64 | 60
Percent change from baseline
  TLC and FRC combined, n = 64, 60 | -6.741 (1.4031) | -7.035 (1.4671)
  TLC, n = 64, 59 | -6.825 (1.4286) | -6.674 (1.5061)
  FRC, n = 64, 60 | -6.494 (1.5027) | -8.281 (1.5752)
Statistical Analysis 1: Comparison: Zemaira® (Early Start) vs Zemaira® (Delayed Start); Analysis of the percent change in lung density (for TLC + FRC combined) from baseline to 2 years was analyzed using an ANCOVA model with country, treatment, and baseline lung density as fixed effects and inspiration state as a repeated random effect; Test type: Superiority or Other; p = 0.883, ANCOVA — Two-sided P-value; Difference in lung density(adjusted P15) = 0.294, 95% CI 2-sided [-3.645 to 4.233]
Statistical Analysis 2: Comparison: Zemaira® (Early Start) vs Zemaira® (Delayed Start); Analysis of the percent change in lung density (for TLC) from baseline to 2 years was analyzed using an ANCOVA model with country, treatment, and baseline lung density as fixed effects; Test type: Superiority or Other; p = 0.941, ANCOVA — Two-sided P-value; Difference in lung density(adjusted P15) = -0.151, 95% CI 2-sided [-4.172 to 3.870]
Statistical Analysis 3: Comparison: Zemaira® (Early Start) vs Zemaira® (Delayed Start); Analysis of the percent change in lung density (for FRC) from baseline to 2 years was analyzed using an ANCOVA model with country, treatment, and baseline lung density as fixed effects; Test type: Superiority or Other; p = 0.404, ANCOVA — Two-sided P-value; Difference in lung density(adjusted P15) = 1.787, 95% CI 2-sided [-2.440 to 6.014]

4. Secondary Outcome: Change in Subject-reported Symptoms
Description: Patient-reported symptoms were measured using the St George's Respiratory Questionnaire (SGRQ). SGRQ total, symptoms, activity and impact scores range from 0 to 100, with higher scores indicating more limitations, and change from baseline below zero (0) is favorable, indicating improvement.
Time Frame: From baseline to 2 years
Population: ITT population. Subjects may not have been included in all efficacy analyses because of missing efficacy assessments.
Measure: Mean (Standard Deviation); unit: units on a scale (change from baseline)
Arm/Group | Zemaira® (Early Start) | Zemaira® (Delayed Start)
Number analyzed (Participants) | 67 | 58
units on a scale (change from baseline)
  Total score, n = 62, 56 | 1.185 (13.624) | 1.499 (12.0507)
  Symptoms score, n = 67, 58 | 6.601 (22.29) | 0.728 (19.2189)
  Activity score, n = 67, 57 | 0.55 (14.1429) | 2.831 (14.0013)
  Impact score, n = 65, 57 | -0.22 (15.8999) | 1.626 (13.5699)

5. Secondary Outcome: Percent Change in Lung Function as Measured by Forced Expiratory Volume in 1 Second (FEV1)
Time Frame: From baseline up to 2 years
Population: ITT population. Subjects may not have been included in all efficacy analyses because of missing efficacy assessments.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Zemaira® (Early Start) | Zemaira® (Delayed Start)
Number analyzed (Participants) | 69 | 56
Percent change from baseline | -8.610 (12.9541) | -8.666 (10.9057)

6. Secondary Outcome: Percent Change in Lung Function as Measured by Ratio of FEV1/FVC (Forced Vital Capacity)
Time Frame: From baseline up to 2 years
Population: ITT population. Subjects may not have been included in all efficacy analyses because of missing efficacy assessments.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Zemaira® (Early Start) | Zemaira® (Delayed Start)
Number analyzed (Participants) | 69 | 56
Percent change from baseline | 0.560 (12.9685) | -5.441 (10.8993)

7. Secondary Outcome: Percent Change in Lung Function as Measured by Percent Predicted FEV1
Time Frame: From baseline up to 2 years
Population: ITT population. Subjects may not have been included in all efficacy analyses because of missing efficacy assessments.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Zemaira® (Early Start) | Zemaira® (Delayed Start)
Number analyzed (Participants) | 68 | 54
Percent change from baseline | -7.165 (13.2053) | -6.958 (11.0846)

8. Secondary Outcome: Number of Subjects With Pulmonary Exacerbations
Time Frame: Up to 2 years
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Zemaira® (Early Start) | Zemaira® (Delayed Start)
Number analyzed (Participants) | 76 | 64
participants
  No exacerbation | 13 | 16
  Overall (at least 1 exacerbation) | 63 | 48
  Moderate exacerbation | 60 | 46
  Severe exacerbation | 17 | 11
  Neither moderate or severe exacerbation | 21 | 17

9. Secondary Outcome: Annual Rate in Subject Years of Pulmonary Exacerbations
Description: Annual exposure-adjusted incidence rate of pulmonary exacerbations.
Time Frame: Up to 2 years
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: Exacerbations/subject year
Arm/Group | Zemaira® (Early Start) | Zemaira® (Delayed Start)
Number analyzed (Participants) | 76 | 64
Exacerbations/subject year | 1.71 [1.49 to 1.92] | 1.39 [1.18 to 1.59]

10. Secondary Outcome: Time to First Pulmonary Exacerbation
Time Frame: Up to 2 years
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Zemaira® (Early Start) | Zemaira® (Delayed Start)
Number analyzed (Participants) | 76 | 64
years | 0.405 [0.315 to 0.687] | 0.602 [0.287 to 0.843]

11. Secondary Outcome: Percentage of Subjects With Treatment Emergent Adverse Events
Description: Percentage of subjects with treatment-emergent adverse events (TEAEs): overall, by severity, by relatedness, by seriousness, and which occurred within 24 hours of Zemaira administration.
Time Frame: From baseline up to 2.5 years
Population: Safety population comprises all subjects who were included in the study and who received at least 1 dose of Zemaira during study CE1226_3001.
Measure: Number; unit: percentage of subjects
Arm/Group | Zemaira® (Early Start) | Zemaira® (Delayed Start)
Number analyzed (Participants) | 76 | 64
percentage of subjects
  Any TEAE | 100 | 96.9
  Mild TEAE | 19.7 | 15.6
  Moderate TEAE | 50.0 | 51.6
  Severe TEAE | 30.3 | 29.7
  Any treatment related TEAE | 14.5 | 10.9
  Any serious TEAE | 36.8 | 35.9
  Any TEAE within 24 hours | 86.8 | 79.7

ADVERSE EVENTS:
Time Frame: Up to 2.5 years
Description: Treatment-emergent adverse events are presented
Groups:
- Zemaira®: The safety population comprised all subjects enrolled in study CE1226_3001 and who received at least 1 administration of Zemaira® during study CE1226_3001.
Arm/Group | Zemaira®
Serious Adverse Events (participants affected / at risk) | 51/140
Other Adverse Events (participants affected / at risk) | 137/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zemaira® (N=140)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 1 (1)
Lung transplant (Surgical and medical procedures) | 1 (1)
Strangulated hernia repair (Surgical and medical procedures) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Palpitations (Cardiac disorders) | 2 (4)
Angina unstable (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 17 (43)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Cerebral thrombosis (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hypotonia (Nervous system disorders) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Condition aggravated (General disorders) | 3 (4)
Chest pain (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2)
Pneumonia (Infections and infestations) | 6 (6)
Lower respiratory tract infection (Infections and infestations) | 4 (8)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 (2)
Anal abscess (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zemaira® (N=140)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 50 (137)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (40)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (27)
Headache (Nervous system disorders) | 28 (58)
Condition aggravated (General disorders) | 27 (71)
Oedema peripheral (General disorders) | 12 (13)
Pyrexia (General disorders) | 10 (15)
Diarrhoea (Gastrointestinal disorders) | 11 (11)
Nausea (Gastrointestinal disorders) | 10 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (19)
Nasopharyngitis (Infections and infestations) | 40 (72)
Lower respiratory tract infection (Infections and infestations) | 20 (106)
Upper respiratory tract infection (Infections and infestations) | 16 (37)
Influenza (Infections and infestations) | 15 (17)
Oral candidiasis (Infections and infestations) | 13 (37)
Bronchitis (Infections and infestations) | 12 (22)
Pneumonia (Infections and infestations) | 10 (17)
Sinusitis (Infections and infestations) | 8 (15)
Urinary tract infection (Infections and infestations) | 8 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.